CLINICAL TRIAL: NCT07024771
Title: A Study On Association Between Neurological Pupil Index and Clinical Severity of Hypoxic Ischemic Encephalopathy In Neonates Admitted To Neonatal Neurocritical Care Unit
Brief Title: Severity of Hypoxic Ischemic Encephalopathy and Neurological Pupil Index in Neonates
Acronym: SHINE
Status: Not yet recruiting | Type: Observational
Sponsor: University of Calgary (Other)
Responsible Party: Sponsor
Other Study IDs: REB25-0010
Record Dates: First submitted 2025-05-22; First posted 2025-06-17 (Actual); Last update posted 2025-06-17 (Actual); Status verified 2025-05

CONDITIONS: Hypoxic Ischemic Encephalopathy (HIE)
Keywords: Neurological pupil index; Hypoxic ischemic encephalopathy; automated pupillometry; neonatal neurocritical care; severity of HIE; therapeutic hypothermia; cooling therapy; NPi; seizures; EEG
MeSH Terms: conditions — Hypoxia-Ischemia, Brain; Seizures

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Device: Yes

GROUPS / COHORTS (1):
- HIE infants: Newborns diagnosed with HIE , more than 35 weeks of age, admitted to a neonatal neurocritical care unit in Alberta Children's hospital, undergoing therapeutic hypothermia
  Interventions: Device: Automated Pupillometer

INTERVENTIONS:
Device: Automated Pupillometer — An automated pupillometer will be used to measure pupil size and calculate NPi in newborns with HIE
  Other Names: Neurological pupil index

SUMMARY:
The goal of this observational study is to learn if the reactivity of a newborn's eye to light (measured as an index, using a new device -pupillometer) reflect the health of their brain recovering from disruption of blood/oxygen supply during birth (Hypoxic Ischemic Encephalopathy-HIE). The main questions it aims to answer are:

* With a decreasing reactivity index, does the chance of an abnormal electrical function of brain (noted by electroencephalography (EEG)) increase?
* With a decreasing reactivity index, do the odds of an indicator of severe impact on brain health (abnormal brain imaging, seizures, feeding difficulty) increase? Participants will undergo eye examination using the pupillometer instead of the regular penlight, as part of their routine neurological examination. This will not change the way in which the newborn is being treated and managed medically.

DETAILED DESCRIPTION:
BACKGROUND:

A newborn baby diagnosed with Hypoxic ischemic encephalopathy (HIE) needs frequent assessment of brain function which includes assessment of pupils in the eyes. However the traditional penlight does not provide a standard measurement and is not very accurate , as it varies based on interpretation of the observer. A new hand-held, non-contact device known as the automated "pupillometer", not only provides a safe, reliable, accurate measurement of the pupil size, but also provides additional information like Neurological Pupil Index (NPi). This value is used to assess the brain function in adults and older children, but the significance of the same has not been studied in a newborn population.

METHODOLOGY:

An Informed consent will be obtained prior to enrolment of the infant in the study. Neurological examination and pupillary assessment will be done at 5 different timepoints: - first at admission(baseline), followed by 24 hours, 48 hours and 72 hours of life, and once prior to discharge. Measurements will be done in both eyes and lesser score of the two will be considered for analysis. Outcome measures including EEG (which is continuous) and MRI (done on day 5 per unit protocol) will be documented and collated for analysis. This is an observational study and the measurement of NPi will not alter the treatment protocol.

The device has been approved by Health Canada for use across all patient population. This device poses no new risks and is safe to use, as it is a non-contact device and is relatively easy to use. Aseptic precautions will be followed when the device is used.

ANALYSIS:

SAMPLE SIZE CONSIDERATIONS:

This is a novel study, with no pre-existing literature. Hence, an initial small scale pilot study will be undertaken with a convenient sample size of all moderate to severe HIE within a year, with anticipation of 70% recruitment. An estimated sample size of 20-25 will help estimate the effect size, variability of NPi, explore relationship between NPi & indicators of severity of HIE and further refine study design & sample size calculation

STATISTICAL ANALYSIS:

Primary outcome:

The primary outcome (abnormal EEG pattern) will be a categorical variable (Yes/No type) The relationship between NPi and the primary outcome will be analysed using logistic regression model and expressed as Odds ratio with 95% confidence intervals.

Secondary outcome:

The secondary outcome (a composite measure of factors which indicate risk for severe HIE (including occurrence of seizure during admission, abnormal MRI finding or persistent feeding difficulty) will be assessed using logistic regression A Receiver-Operator Characteristic curve analysis will evaluate the diagnostic accuracy of NPi in predicting clinical severity of HIE indicating sensitivity & specificity. Any novel threshold values which can predict the cut-off for abnormal EEG pattern, or risk of severe HIE using other indicators will be identified with AUC >0.7

ELIGIBILITY:
Inclusion Criteria:

* Neonates ≥35 weeks of GA, with Hypoxic ischemic encephalopathy admitted to neonatal neuro-intensive care unit at Alberta children's hospital, Calgary will be included in the study

Exclusion Criteria:

* Infants with chromosomal abnormalities/ syndromic associations
* Infants with ocular / orbital injuries or structural anomalies of the eye obscuring the pupillometry measurement
* Infants with inadequate pupillometry data / EEG data

Max Age: 6 Hours | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Neonates ≥35 weeks of GA, with Hypoxic ischemic encephalopathy admitted to neonatal neuro-intensive care unit at Alberta children's hospital, Calgary
Sampling Method: Non-Probability Sample
Enrollment: 25 (Estimated)
Dates: Start 2025-08 (Estimated); Primary Completion 2026-06 (Estimated); Study Completion 2026-06 (Estimated)

PRIMARY OUTCOMES:
Abnormal EEG pattern | From starting therapeutic hypothermia at admission (baseline) till completion of therapeutic hypothermia (72 hours from starting cooling therapy). EEG will be monitored CONTINUOUSLY during this period of 72 hours
  Abnormal EEG patterns will be monitored via continuous amplitude -integrated EEG (aEEG) . It will be scored by an expert neonatal neurologist into an objective score ranging from 0 to 5, where 0 = normal, 1=discontinuous, 2= Burst suppression, 3= isoelectric, 4= seizures and 5= not done. Any score from 1 to 4 will be considered as indicative of severe HIE, and will be considered collectively as "abnormal EEG pattern"

SECONDARY OUTCOMES:
Abnormal MRI findings | MRI brain will be done and scored between day 4 and day 5 from admission
  To identify any association between NPi and abnormal MRI brain findings
  * MRI brain findings will be interpreted by an expert neuro-radiologist and classified based on modified WEEKE's score;
  * any score >3 will be considered abnormal and indicate severe HIE
Presence of seizure | baseline (day of admission) till day 5 after admission
  To identify any association between NPi and occurrence of seizure during the hospital stay.
  -Occurrence of seizure during the hospital stay will be monitored for and documented as YES/NO response based on presence or absence of seizure activity
persistent Feeding difficulty | will be assessed at the time of discharge from NICU to home or transfer to ward (anytime between week 1 to week 4)
  To identify any association between NPi and persistent feeding difficulty at discharge.
  * Persistent feeding difficulty will be defined as requiring tube feeds / home gavage feeds at the time of discharge
  * will be documented as YES/NO response based on presence or absence of feeding difficulty

CONTACTS AND LOCATIONS:
Overall Officials: Khorshid Mohammad, MD, MSc, FRCP, FRCPC, Principal Investigator — Cummings school of medicine, University of Calgary
Locations (1):
- University of Calgary, Calgary, Alberta, Canada

IPD SHARING:
Plan to Share IPD: No
per data sharing restrictions , considering confidentiality of information, in a vulnerable population, IPD will not be shared

REFERENCES:
- [Background] Oddo M, Sandroni C, Citerio G, Miroz JP, Horn J, Rundgren M, Cariou A, Payen JF, Storm C, Stammet P, Taccone FS. Quantitative versus standard pupillary light reflex for early prognostication in comatose cardiac arrest patients: an international prospective multicenter double-blinded study. Intensive Care Med. 2018 Dec;44(12):2102-2111. doi: 10.1007/s00134-018-5448-6. Epub 2018 Nov 26. PMID 30478620
- [Background] Riker RR, Sawyer ME, Fischman VG, May T, Lord C, Eldridge A, Seder DB. Neurological Pupil Index and Pupillary Light Reflex by Pupillometry Predict Outcome Early After Cardiac Arrest. Neurocrit Care. 2020 Feb;32(1):152-161. doi: 10.1007/s12028-019-00717-4. PMID 31069659
- [Background] Al-Obaidi SZ, Atem FD, Stutzman SE, Olson DM. Impact of Increased Intracranial Pressure on Pupillometry: A Replication Study. Crit Care Explor. 2019 Oct 30;1(10):e0054. doi: 10.1097/CCE.0000000000000054. eCollection 2019 Oct. PMID 32166235
- [Background] Kim TJ, Park SH, Jeong HB, Ha EJ, Cho WS, Kang HS, Kim JE, Ko SB. Neurological Pupil Index as an Indicator of Neurological Worsening in Large Hemispheric Strokes. Neurocrit Care. 2020 Oct;33(2):575-581. doi: 10.1007/s12028-020-00936-0. PMID 32096118
- [Background] Shah SS, Ranaivo HR, Mets-Halgrimson RB, Rychlik K, Kurup SP. Establishing a normative database for quantitative pupillometry in the pediatric population. BMC Ophthalmol. 2020 Mar 26;20(1):121. doi: 10.1186/s12886-020-01389-x. PMID 32216772
- [Background] Sandroni C, Citerio G, Taccone FS. Automated pupillometry in intensive care. Intensive Care Med. 2022 Oct;48(10):1467-1470. doi: 10.1007/s00134-022-06772-4. Epub 2022 Jun 30. No abstract available. PMID 35773500
- [Background] Jiang J, Sari H, Goldman R, Huff E, Hanna A, Samraj R, Gourabathini H, Bhalala U. Neurological Pupillary Index (NPi) Measurement Using Pupillometry and Outcomes in Critically Ill Children. Cureus. 2023 Oct 4;15(10):e46480. doi: 10.7759/cureus.46480. eCollection 2023 Oct. PMID 37927706
- [Background] Couret D, Boumaza D, Grisotto C, Triglia T, Pellegrini L, Ocquidant P, Bruder NJ, Velly LJ. Reliability of standard pupillometry practice in neurocritical care: an observational, double-blinded study. Crit Care. 2016 Mar 13;20:99. doi: 10.1186/s13054-016-1239-z. PMID 27072310
- [Background] Hall CA, Chilcott RP. Eyeing up the Future of the Pupillary Light Reflex in Neurodiagnostics. Diagnostics (Basel). 2018 Mar 13;8(1):19. doi: 10.3390/diagnostics8010019. PMID 29534018
- [Background] Brown KL, Agrawal S, Kirschen MP, Traube C, Topjian A, Pressler R, Hahn CD, Scholefield BR, Kanthimathinathan HK, Hoskote A, D'Arco F, Bembea M, Manning JC, Hunfeld M, Buysse C, Tasker RC. The brain in pediatric critical care: unique aspects of assessment, monitoring, investigations, and follow-up. Intensive Care Med. 2022 May;48(5):535-547. doi: 10.1007/s00134-022-06683-4. Epub 2022 Apr 21. PMID 35445823
- [Background] van Kooij BJ, van Handel M, Nievelstein RA, Groenendaal F, Jongmans MJ, de Vries LS. Serial MRI and neurodevelopmental outcome in 9- to 10-year-old children with neonatal encephalopathy. J Pediatr. 2010 Aug;157(2):221-227.e2. doi: 10.1016/j.jpeds.2010.02.016. Epub 2010 Apr 9. PMID 20381069
- [Background] Hagberg H, David Edwards A, Groenendaal F. Perinatal brain damage: The term infant. Neurobiol Dis. 2016 Aug;92(Pt A):102-12. doi: 10.1016/j.nbd.2015.09.011. Epub 2015 Sep 25. PMID 26409031
- See also: NeurOptics: NPI-200 Pupillometer. Instructions for use . (2021). — https://neuroptics.com/wp-content/uploads/2017/02/NPi-200_Instructions.pdf